CLINICAL TRIAL: NCT06277050
Title: Maintenance Therapy With Toripalimab Combined With Capecitabine Versus Maintenancetherapy With Capecitabine Alone in High-risk Nasopharyngeal Carcinoma: a Multicenter, Prospective, Randomized Phase III Clinical Trial (NPC-ICMB)
Brief Title: Maintenance Therapy With Toripalimab and Capecitabine Versus Capecitabine Alone in High-risk Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC-ICMB
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-02

CONDITIONS: Nasopharyngeal Carcinoma; High-Risk Cancer; Maintenance Therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Maintenance; toripalimab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintenance Therapy with Toripalimab and Capecitabine (Experimental): Capecitabine maintenance therapy (1000 mg/m2 orally twice daily on days 1-14) every 3 weeks. Maintenance therapy of Toripalimab (240 mg, every 3 weeks). The total treatment time of oral chemotherapy is 12 months.
  Interventions: Drug: Maintenance Therapy with Toripalimab and Capecitabine
- Maintenance Therapy with Capecitabine alone (Active Comparator): Capecitabine maintenance therapy (1000 mg/m2 orally twice daily on days 1-14) every 3 weeks. The total treatment time of oral chemotherapy is 12 months.
  Interventions: Drug: Maintenance Therapy with Capecitabine

INTERVENTIONS:
Drug: Maintenance Therapy with Toripalimab and Capecitabine — Capecitabine maintenance therapy (1000 mg/m2 orally twice daily on days 1-14) every 3 weeks. Maintenance therapy of Toripalimab (240 mg, every 3 weeks). The total treatment time of oral chemotherapy is 12 months.
  Arms: Maintenance Therapy with Toripalimab and Capecitabine
Drug: Maintenance Therapy with Capecitabine — Capecitabine maintenance therapy (1000 mg/m2 orally twice daily on days 1-14) every 3 weeks. The total treatment time of oral chemotherapy is 12 months.
  Arms: Maintenance Therapy with Capecitabine alone

SUMMARY:
N3 classification, rENE positivity is a high-risk type of locally advanced nasopharyngeal carcinoma. EBV DNA remaining at detectable levels after induction chemotherapy is also a characteristic of high-risk nasopharyngeal carcinoma. Based on the available evidence, patients with high-risk nasopharyngeal carcinoma are recommended to receive oral maintenance therapy to reduce the risk of failure.

The purpose of this study was to conduct a prospective, multicenter, randomized phase III clinical trial to determine whether maintenance therapy with triprilimab combined with capecitabine is better than maintenance therapy with capecitabine alone in high-risk nasopharyngeal carcinoma (N3+, rENE+, Detectable EBV DNA after 2 cycles of induction chemotherapy).

DETAILED DESCRIPTION:
The study randomly divided these three types of high-risk nasopharyngeal carcinoma into two groups. The experimental group received maintenance therapy with toripalimab and capecitabine, while the control group received maintenance therapy with capecitabine alone. The maintenance treatment period of the two groups was 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed nasopharyngeal carcinoma;
2. High-risk nasopharyngeal cancer meets one of three points: a. TanyN3M0; b. High-grade rENE, coalescent nodal or invasion of surrounding structures (muscle, skin, nerves, etc.); c. Detectable EBV DNA after 2 cycles of induction chemotherapy.

3.18-70 years old, both genders; 4. ECOG≤1; 5. Received 2-3 cycles of induction chemotherapy and concurrent chemoradiotherapy (intensity-modulated radiotherapy); 6. Patients must have adequate organ function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment) as determined by: Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ 75×109/L; Hemoglobin ≥ 9 g/dL; serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN), (for subjects with liver metastases, TBIL ≤3×ULN; ALT and AST≤5×ULN); Creatinine ≤1.5×ULN or creatinine clearance rate≥50 ml/min (Cockcroft-Gault formula); serum albumin ≥28 g/L.

7. All women with fertility potential must undergo a urine or serum pregnancy test during screening and the results are negative; 8. Written informed consent;

Exclusion Criteria:

1. Recurrent or distant metastatic nasopharyngeal carcinoma.
2. History of malignant tumors (except cured basal cell carcinoma or uterine cervical carcinoma in situ) within the last 5 years.
3. Has received any prior radiotherapy (RT) or systemic anti-cancer therapy including investigational agents for NPC
4. Has received prior therapy with an anti-PD-1 mab.
5. Active autoimmune diseases or history of autoimmune diseases that may relapse.

   Note: Patients with the following diseases are not excluded and may proceed to further screening:
   1. Controlled Type I diabetes
   2. Hypothyroidism (provided it is managed with hormone replacement therapy only)
   3. Controlled celiac disease
   4. Skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, alopecia) Any other disease that is not expected to recur in the absence of external triggering factors.
6. Any condition that required systemic treatment with either corticosteroids (>10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤14 days before the start of the study。

   Note: Patients who are currently or have previously been on any of the following steroid regimens are not excluded:
   1. Adrenal replacement steroid (dose ≤10 mg daily of prednisone or equivalent)
   2. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption
   3. Short course (≤7 days) of corticosteroid prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a non-autoimmune condition (e.g., delayed-type hypersensitivity reaction caused by contact allergen)。
7. With history of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.
8. With severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc.

   1. Severe infections within 4 weeks before the start of the study, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
   2. Received therapeutic oral or intravenous antibiotics within 2 weeks before start of the study.
9. A known history of HIV infection
10. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers whose HBV DNA is >1000 IU/mL or patients with active hepatitis C virus (HCV) should be excluded. Note: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA <1000 IU/mL), and cured hepatitis C patients can be enrolled.
11. Any major surgical procedure requiring general anaesthesia ≤28 days before start of study。
12. Prior allogeneic stem cell transplantation or organ transplantation.
13. Any of the following cardiovascular risk factors:

    1. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤28 days before start of study
    2. Pulmonary embolism ≤28 days before start of study
    3. Any history of acute myocardial infarction ≤6 months before start of study
    4. Any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV ≤6 months before start of study
    5. Any event of ventricular arrhythmia ≥Grade 2 in severity ≤6 months before start of study
    6. Any history of cerebrovascular accident ≤6 months before start of study
    7. Uncontrolled hypertension: systolic pressure ≥160 mmHg or diastolic pressure ≥100 mmHg despite anti-hypertension medications ≤28 days before start of study
    8. Any episode of syncope or seizure ≤28 days before start of study.
14. A history of severe hypersensitivity reactions to toripalimab, capecitabine and/or any of its excipients.
15. Has received any herbal medicine used to control cancer within 14 days of the start of study
16. Patients with toxicities (as a result of prior anticancer therapy) which have not recovered to baseline or stabilized, except for AEs not considered a likely safety risk (e.g., alopecia, neuropathy and specific laboratory abnormalities)
17. Concurrent participation in another therapeutic clinical study
18. Emotional disturbance or mental illness
19. Refusal or inability to sign informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2029-02-20 (Estimated); Study Completion 2030-02-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 3 years
  Time from date of start of treatment to disease progression or death from any cause.

SECONDARY OUTCOMES:
Distant Metastasis-Free Survival | 3 years
  Time from date of start of treatment to documented distant metastasis or death from any cause, patients with locoregional relapse as a first event will be censored at date of locoregional relapse.
Overall Survival | 3 years
  Time from date of start of treatment to death from any cause, where patients lost to follow-up were censored at the date of last follow-up.
Loco-Regional Recurrence-Free Survival | 3 years
  Time from date start of treatment to documented locoregional relapse or death from any cause, patients with distant metastasis as a first event will be censored at the date of distant metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Jingao Li, Study Chair — Jiangxi Provincial Cancer Hospital
Locations (3):
- China (3):
  - Ganzhou Cancer Hospital, Ganzhou, Jiangxi
  - First Affiliated hospital of Gannan Medical University, Guangzhou, Jiangxi
  - Department of Nasopharyngeal Carcinoma, Jiangxi Cancer Hospital, Nanchang, None Selected

IPD SHARING:
Plan to Share IPD: No